CLINICAL TRIAL: NCT03205046
Title: A Phase 1/2 Proof-of-Concept Study of the Combination of Acalabrutinib and Vistusertib in Subjects With Relapsed/Refractory B-cell Malignancies
Brief Title: A Study of Acalabrutinib and Vistusertib in Subjects With Relapsed/Refractory B-cell Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision not to pursue further development of the combination in DLBCL
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-LY-110
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: DLBCL; Richter Syndrome
MeSH Terms: interventions — acalabrutinib; vistusertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 continuous dose for vistusertib (Experimental): acalabrutinib daily + vistusertib daily
  Interventions: Drug: acalabrutinib; Drug: vistusertib
- Part 1 intermittent dose for vistusertib (Experimental): acalabrutinib daily + vistusertib 5 days on and 2 days off
  Interventions: Drug: acalabrutinib; Drug: vistusertib

INTERVENTIONS:
Drug: acalabrutinib — Acalabrutinib is a selective, irreversible small molecule Bruton's tyrosine kinase (BTK) inhibitor.
  Other Names: ACP-196
Drug: vistusertib — Vistusertib is an inhibitor of mechanistic target of rapamycin (mTOR) kinase
  Other Names: AZD2014

SUMMARY:
This study evaluates the safety of acalabrutinib and vistusertib when taken in combination.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsed/refractory diffuse large B-cell lymphoma (DLBCL) as documented by medical records and with histology based on criteria established by The World Health Organization (WHO):

   * If a subject has de novo DLBCL, the diagnosis is confirmed by biopsy and is immunohistologically characterized as de novo germinal center B-cell-like (GCB) DLBCL or de novo non-GCB DLBCL.
   * If the subjects has Richter's Syndrome (RS), the diagnosis is confirmed by biopsy and is immunohistologically characterized as transformation to DLBCL.
   * If the subjects has transformed DLBCL, the diagnosis is confirmed by biopsy and is immunohistologically characterized as transformation to DLBCL from indolent lymphoma (eg, follicular lymphoma).
2. Men and women ≥18 years of age.
3. Prior treatment for lymphoid malignancy:

   * If the subject has DLBCL, there is no curative option with conventional therapy and the prior treatment included ≥ 1 prior combination chemoimmunotherapy regimen.
   * If the subject has RS, the subject must have had ≥1 prior treatment with a combination chemoimmunotherapy regimen.
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
5. Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of a ≥1.5 cm lesion, as measured in the longest dimension by computed tomography [CT] scan).

Exclusion Criteria:

1. As judged by the Investigator, any evidence of severe or uncontrolled systemic disease (eg, severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease]), or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension, history of, or active, bleeding diatheses (eg, hemophilia or von Willebrand disease) or uncontrolled active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment), or intravenous anti-infective treatment within 2 weeks before first dose of study drug.
2. Diagnosis of PMBCL.
3. Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal (GI) function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
4. History of central nervous system (CNS) lymphoma, leptomeningeal disease or spinal cord compression.
5. Any clinically significant pre-existing severe renal disease (eg, glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis) or high risk of developing severe renal impairment.
6. Abnormal echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) at baseline (left ventricular ejection fraction [LVEF] <40% and shortening fraction <15%). Appropriate correction to be used, if a MUGA is performed.
7. Mean resting corrected QT interval (QTc) calculated using Fridericia's formula (QTcF) >450 msec obtained from 3 electrocardiograms (ECGs); family or personal history of long or short QT syndrome; Brugada syndrome or known history of QTc prolongation or torsade de pointes within 12 months of the subject entering the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (11):
- United States (7):
  - Research Site, Fairway, Kansas
  - Research Site, Bethesda, Maryland
  - Research Site, Rochester, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Hackensack, New Jersey
  - Research Site, Nashville, Tennessee
  - Research Site, Seattle, Washington
- United Kingdom (4):
  - Research Site, Headington
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Collins GP, Clevenger TN, Burke KA, Yang B, MacDonald A, Cunningham D, Fox CP, Goy A, Gribben J, Nowakowski GS, Roschewski M, Vose JM, Vallurupalli A, Cheung J, Raymond A, Nuttall B, Stetson D, Dougherty BA, Schalkwijk S, Carnevalli LS, Willis B, Tao L, Harrington EA, Hamdy A, Izumi R, Pease JE, Frigault MM, Flinn I. A phase 1/2 study of the combination of acalabrutinib and vistusertib in patients with relapsed/refractory B-cell malignancies. Leuk Lymphoma. 2021 Nov;62(11):2625-2636. doi: 10.1080/10428194.2021.1938027. Epub 2021 Jul 16. PMID 34269152
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-110&attachmentIdentifier=ad5df82e-668e-4472-8aac-b20b8fd83f17&fileName=D2276C00002_(ACE-LY-110)_Protocol_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-110&attachmentIdentifier=6cbe6bde-57cb-4e13-b71a-8091a71e3412&fileName=D2276C00002_(ACE-LY-110)_Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Acalabrutinib 100 mg BID Plus Vistusertib BID Continuous: Acalabrutinib daily + Vistusertib daily over the 28-day cycle
- Acalabrutinib 100 mg BID Plus Vistusertib BID Intermittent: Acalabrutinib daily + Vistusertib 2 days on/ 5 days off over the 28-day cycle
Period: Overall Study
Arm/Group | Acalabrutinib 100 mg BID Plus Vistusertib BID Continuous | Acalabrutinib 100 mg BID Plus Vistusertib BID Intermittent
Started | 13 | 12
Completed | 0 | 2
Not Completed | 13 | 10
Not completed — Death | 10 | 6
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study terminated by sponsor | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Acalabrutinib 100 mg BID* Plus Vistusertib BID* Continuous: Acalabrutinib daily + Vistusertib daily over the 28-day cycle
- Acalabrutinib 100 mg BID* Plus Vistusertib BID* Intermittent: Acalabrutinib daily + Vistusertib 2 days on/ 5 days off over the 28-day cycle
- Total: Total of all reporting groups
Arm/Group | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Continuous | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Intermittent | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (15.9) | 67.3 (12.0) | 65.4 (13.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 9 | 14
  United Kingdom | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs)
Description: Safety assessments comprised type, frequency, severity, and relationship to either or both study drug of any AEs or abnormalities of laboratory tests; serious adverse events (SAEs); dose-limiting toxicities (DLTs); or AEs that led to dose modification, dose delay, or discontinuation of study drug(s).
Time Frame: From first dose of study drug until 30 days post last dose
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Continuous | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Intermittent
Number analyzed (Participants) | 13 | 12
Participants | 13 | 12

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Other Adverse Events were assessed from first dose of study drug until 30 days post last dose; All-Cause Mortality was assessed from first dose of study drug until death, loss to follow up, sponsor decision to stop trial, or withdrawal of consent, whichever occurred first, an average of approximately 6 months.
Arm/Group | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Continuous | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Intermittent
All-Cause Mortality (participants affected / at risk) | 10/13 | 6/12
Serious Adverse Events (participants affected / at risk) | 2/13 | 6/12
Other Adverse Events (participants affected / at risk) | 13/13 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Continuous (N=13) | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Intermittent (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Computerised tomogram thorax abnormal (Investigations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Continuous (N=13) | Acalabrutinib 100 mg BID* Plus Vistusertib BID* Intermittent (N=12)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (7)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (7)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (13)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 2 (5)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 8 (10)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 5 (6)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 8 (10)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (4)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 4 (5) | 7 (11)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 2 (2)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (3)
Platelet count decreased (Investigations) | 1 (1) | 1 (3)
Weight decreased (Investigations) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (5) | 5 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (6)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (3)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 5 (6)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment to this study was stopped early by the sponsor and an abbreviated CSR was generated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT03205046/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT03205046/SAP_001.pdf